CLINICAL TRIAL: NCT05477472
Title: Observational Study of the Efficacy and Tolerability of Low-dose Phytotherapy Using the Example of St John's Wort (Hypericum Perforatum)
Brief Title: Low Dose St John's Wort for Depression
Status: Completed | Type: Observational
Sponsor: Ceres Heilmittel AG (Industry)
Collaborators: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: OS01
Record Dates: First submitted 2022-06-27; First posted 2022-07-28 (Actual); Last update posted 2022-07-28 (Actual); Status verified 2022-07

CONDITIONS: Major Depression
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Hypericum extract LI 160

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: St John's Wort — daily intake of CERES St John's Wort mother tincture. Dose according to the treating physician.
  Other Names: CERES St John's Wort mother tincture

SUMMARY:
This observational study observes the routine use of low-dose St John's Wort herbal mother tincture in patients with major depression. It measures intensity of depression at the beginning of St Johns Wort and after 6 weeks and evaluates tolerability and compliance.

DETAILED DESCRIPTION:
Herbal medicine is widely used, and high-quality evidence shows their efficacy and tolerability for specific disorders. Most of the studies, however, is conducted with standardized, relatively high dosed dry extract preparations, while other preparations such as tinctures are widely used as well. The aim of this observational study ist to document real-live use of the use of a low-dose herbal medicine preparation (a mother tincture) of St John's Wort (Hypericum perforatum), to compare depression intensity at the beginning and after 6 weeks of therapy using the Hamilton Depression Scale 17, and to evaluate tolerability and compliance. Finally, the results will be compared with results of randomized controlled trials examining high dosed dry extract preparations of St John's Wort for major depression.

ELIGIBILITY:
Inclusion Criteria:

* diagnosis of mild or moderate depression according to ICD-10 or DSM-IV
* new start of CERES St John's wort mother tincture

Exclusion Criteria:

- at the same time as St John's wort mother tincture started, other antidepressive therapy

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: patients of outpatient physicians which are used to the therapy of major depression with CERES St John's Wort mother tincture
Sampling Method: Non-Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2005-08 (Actual); Primary Completion 2007-01 (Actual); Study Completion 2007-01 (Actual)

PRIMARY OUTCOMES:
Hamilton Depression Scale 17 | Change at 6 weeks
  validated tool to measure depression intensity. Maximum score 51, minimum 0. Higher score means higher intensity of depressive symptoms.

CONTACTS AND LOCATIONS:
Overall Officials: Natalie Kalbermatten, cand. med., Principal Investigator — University of Zurich
Locations (1):
- CERES Heilmittel AG, Kesswil, Thurgau, Switzerland

IPD SHARING:
Plan to Share IPD: No